CLINICAL TRIAL: NCT02832960
Title: Impact of Thyroid Hormone Replacement on Cardiac Function: a Randomized Placebo-Controlled Trial in Older Adults With Subclinical Hypothyroidism
Brief Title: The TRUST Trial - CardioVascular Imaging ECHO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Lausanne Hospitals (Other); University Hospital, Geneva (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 162/11_4; 974a (Other Grant/Funding Number: VELUX STIFTUNG)
Record Dates: First submitted 2016-07-12; First posted 2016-07-14 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Thyroid Dysfunction; Atherosclerosis; Heart Failure
Keywords: Thyroid Dysfunction; Atherosclerosis; Heart Failure; Cardiovascular imaging; Randomized Controlled Trial
MeSH Terms: conditions — Atherosclerosis; Heart Failure | interventions — Thyroxine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): The intervention will start with Levothyroxine 50 mcg daily (reduced to 25 mcg in subjects <50 kg of body weight or if known coronary heart disease - previous myocardial infarction or symptoms of angina pectoris) vs. matching placebo; at 3 months, if the serum TSH level is <0.4 mU/L, dose will be reduced by 25 mcg; TSH >=0.4 and <4.6 mU/L, no change to dose; TSH >=4.6 mU/L, additional 25 mcg. The process will be repeated at 12 months, then annually; mock titration will be performed in the placebo group. The maximum possible dose of Levothyroxine which will be prescribed is 150 mcg (after 4 increments of 25 mcg at 3 months, 1, 2, 3 years; from the starting dose of 50 mcg).
  Interventions: Drug: Levothyroxine
- 2 (Placebo Comparator): Control patients will obtain a placebo pill of the same characteristics as the intervention drug, and mock titration will be carried out identically to the intervention drug. Pharmaceutical composition of placebo (100 mg): Lactose monohydrate 66 mg, Maize starch 25 mg, Gelatin 5 mg, Croscarmellose sodium 3.5 mg, Magnesium stearate (vegetable source) 0.5 mg.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levothyroxine — The intervention will start with Levothyroxine 50 mcg daily (reduced to 25 mcg in subjects <50 kg of body weight or if known coronary heart disease - previous myocardial infarction or symptoms of angina pectoris) vs. matching placebo; at 3 months, if the serum TSH level is <0.4 mU/L, dose will be reduced by 25 mcg; TSH >=0.4 and <4.6 mU/L, no change to dose; TSH >=4.6 mU/L, additional 25 mcg. The process will be repeated at 12 months, then annually; mock titration will be performed in the placebo group. The maximum possible dose of Levothyroxine which will be prescribed is 150 mcg (after 4 increments of 25 mcg at 3 months, 1, 2, 3 years; from the starting dose of 50 mcg).
  Arms: 1
Drug: Placebo — Control patients will obtain a placebo pill of the same characteristics as the intervention drug, and mock titration will be carried out identically to the intervention drug. Pharmaceutical composition of placebo (100 mg): Lactose monohydrate 66 mg, Maize starch 25 mg, Gelatin 5 mg, Croscarmellose sodium 3.5 mg, Magnesium stearate (vegetable source) 0.5 mg.
  Arms: 2

SUMMARY:
Coronary heart disease (CHD) and heart failure (HF) are the leading causes of mortality and morbidity, particularly with the current context of an aging population. Prospective cohort studies, as well as analyses of pooled individual participant data suggest up to a 60-90% increase in the risk of CHD or HF events among adults with severe SHypo. However, no large randomized controlled trials (RCT) have assessed the impact of thyroid replacement on cardiovascular (CV) imaging outcomes. The goals of this proposal are to address the impact of thyroid replacement on cardiac function. The investigators will conduct a RCT in 185 patients with subclinical hypothyroidism who will be randomly assigned to thyroxine or placebo with an average follow-up of 24 months from baseline. The main outcome will be CV imaging modalities measured by echocardiography at the close-out visit. Assessment of the impact of thyroid replacement on cardiac function and subclinical atherosclerosis within a trial will aid decisions and evidence-based guidelines development to treat a potential modifiable risk factor, such as SHypo.

DETAILED DESCRIPTION:
Background: Coronary heart disease (CHD) and heart failure (HF) are the leading causes of mortality and morbidity, particularly with the current context of an aging population. Subclinical hypothyroidism (SHypo), defined as elevated serum TSH levels with normal thyroxine values, is common in older adults (5-10%). Prospective cohort studies, as well as analyses of pooled individual participant data suggest up to a 60-90% increase in the risk of CHD or HF events among adults with severe SHypo. However, no large randomized controlled trials (RCT) have assessed the impact of thyroid replacement on cardiovascular (CV) imaging outcomes (largest trial to date: 45 participants). Imaging endpoints are especially well-suited for early trials with investigational therapies for HF treatment and prevention, as well as validated and strong surrogate markers of clinical outcomes.

Specific Aims: The goals of this proposal are to address the impact of thyroid replacement on 1) cardiac function as measured by echocardiography.

Methods: The investigators will conduct a RCT in 185 patients with subclinical hypothyroidism who will be randomly assigned to thyroxine or placebo with an average follow-up of 24 months from baseline (4 death and 17 withdrawal). The main outcome will be CV imaging modalities measured by echocardiography at the close-out visit. Transthoracic echocardiography will be performed for the assessment of diastolic function (abnormalities of the pulsed wave mitral valve inflow pattern and mitral annulus tissue velocities, left atrial volume index, left ventricular [LV] mass index) and cardiac systolic function (LV ejection fraction and regional function). Ultrasound of carotid intima media thickness (CIMT) will be used to assess subclinical atherosclerosis and plaque burden. All images will be centralized at the core lab for a blinded and standardized interpretation.

Expected value of the proposed project: Controversies persist regarding the indications for screening and treatment of SHypo due to the lack of an appropriately powered RCT addressing the impact of thyroid replacement on CV outcomes. Assessment of the impact of thyroid replacement on cardiac function and subclinical atherosclerosis within a trial will aid decisions and evidence-based guidelines development to treat a potential modifiable risk factor, such as SHypo. The strengths of this study include the combination of: 1) High feasibility of the project in collaboration with the largest RCT on SHypo making it possible to investigate the mechanisms of associations with CV disease; 2) Innovative project with combined CV imaging to assess cardiac function with thyroid replacement therapy vs. placebo; 3) Excellent power given the large sample size and participants' older age. The sample size for this proposal will be 5-fold higher than previous small trials of thyroid replacement on CV outcomes. The collaboration of CV imaging modalities expertise with the ongoing largest trial on SHypo, is a unique opportunity to address the clinical and scientific issue of the impact of SHypo on the CV system.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling patients aged >= 65 years with subclinical hypothyroidism
* Written informed consent

Exclusion Criteria:

* Subjects currently under levothyroxine or antithyroid drugs (amiodarone, lithium)
* Recent thyroid surgery or radio-iodine (within 12 months)
* Grade IV NYHA heart failure
* Prior clinical diagnosis of dementia
* Recent hospitalization for major illness or elective surgery (within 4 weeks)
* Terminal illness
* Patients with rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption
* Subjects who are participating in ongoing RCTs of therapeutic interventions (including CTIMPs)
* Plan to move out of the region in which the trial is being conducted within the next 2 years (proposed minimum follow-up period)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 185 (Actual)
Dates: Start 2016-06; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Diastolic cardiac Function as measured by echocardiography | one year follow up
Systolic cardiac Function as measured by echocardiography | one year follow up

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Rodondi, MD MAS, Principal Investigator — University Clinic of General Internal Medicine, Bern University Hospital, Bern
Locations (3):
- Switzerland (3):
  - Cardiology Division, Geneva University Hospitals, Geneva, Canton of Geneva
  - Department of General Internal Medicine, Lausanne, Canton of Vaud
  - Clinic for General Internal Medicine, Bern University Hospital Bern, Bern

REFERENCES:
- [Background] Rodondi N, den Elzen WP, Bauer DC, Cappola AR, Razvi S, Walsh JP, Asvold BO, Iervasi G, Imaizumi M, Collet TH, Bremner A, Maisonneuve P, Sgarbi JA, Khaw KT, Vanderpump MP, Newman AB, Cornuz J, Franklyn JA, Westendorp RG, Vittinghoff E, Gussekloo J; Thyroid Studies Collaboration. Subclinical hypothyroidism and the risk of coronary heart disease and mortality. JAMA. 2010 Sep 22;304(12):1365-74. doi: 10.1001/jama.2010.1361. PMID 20858880
- [Background] Gencer B, Collet TH, Virgini V, Bauer DC, Gussekloo J, Cappola AR, Nanchen D, den Elzen WP, Balmer P, Luben RN, Iacoviello M, Triggiani V, Cornuz J, Newman AB, Khaw KT, Jukema JW, Westendorp RG, Vittinghoff E, Aujesky D, Rodondi N; Thyroid Studies Collaboration. Subclinical thyroid dysfunction and the risk of heart failure events: an individual participant data analysis from 6 prospective cohorts. Circulation. 2012 Aug 28;126(9):1040-9. doi: 10.1161/CIRCULATIONAHA.112.096024. Epub 2012 Jul 19. PMID 22821943